CLINICAL TRIAL: NCT04674696
Title: Phase II Study of Short-course Radiotherapy With Induction and Consolidation Chemotherapy in Patients With Locally Advanced High-risk Rectal Cancer
Brief Title: Short-course Radiotherapy With Induction and Consolidation Chemotherapy in Patients With Locally Advanced Rectal Cancer
Acronym: SHORT-ICAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto Nacional de Cancer, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHORT-ICAR
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-11

CONDITIONS: Rectal Cancer; Total Neoadjuvant Treatment
Keywords: rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): Patients will receive 2 CAPOX cycles, followed by short-course radiotherapy and 4 CAPOX cycles.
  Interventions: Other: Approach

INTERVENTIONS:
Other: Approach — Patients will receive 2 CAPOX cycles, followed by short-course radiotherapy and 4 CAPOX cycles.

SUMMARY:
Short-course radiotherapy followed by consolidation chemotherapy has shown a better response rate when compared to chemoradiotherapy treatment.

In addition, recent studies have shown better tolerance with total neoadjuvant treatment, with induction or consolidation chemotherapy. Induction chemotherapy could reduce the size of the tumor, treat micrometastases early and allow treatment to start immediately (avoiding potential delays in waiting for radiotherapy). While consolidation chemotherapy allows longer waiting times for surgery, with higher response rates.

DETAILED DESCRIPTION:
Methods: This trial aim to evaluate induction treatment with CAPOX, followed by short-course radiotherapy consolidation chemotherapy with CAPOX. After 5-7 weeks, patients will be evaluate by MRI. Patients with incomplete clinical response will be referred to immediate surgery and patients with complete clinical response will be managed with "watch and wait" approach. Patients with progression disease during the treatment phase will be withdrawn from the study and will receive their treatment according to the investigator's judgment.

The sample size was calculated according to Simon's optimal two-stage design. Accordingly, 21 patients must be included in each group during the first stage and 24 during the second stage. Treatment regimen will be considered effective if 9 or more patients show good response (final analysis), reaching 80% power with an alpha of 0.10 level of significance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of mid or low rectum
* Locally advanced rectal cancer with one of the high-risk factors confirmed by high-resolution thin-slice Magnetic resonance image (3 mm) tumors extending to within 1 mm of, or beyond the mesorectal fascia; tumor extending 5 mm or more into perirectal fat; resectable cT4 tumors; lower third; nodal involvement; extramural vascular invasion
* ECOG performance status of 0-2
* An informed consent has been signed by the patient

Exclusion Criteria:

* Upper rectal cancer
* Metastatic disease
* The patient received any previous therapy for colorectal cancer or another malignancy
* Other malignant tumours within the last 5 years except cervical carcinoma in situ and basal cell carcinoma of the skin
* Previous thromboembolic or haemorrhagic events within 6 months prior to registration
* Patients with malabsorption syndrome or difficulties in swallowing
* The patient has severe underlying diseases or poor condition to receive chemotherapy or radiotherapy
* Pregnant of breastfeeding women
* The patient who participate in another clinical trial, or receives any drug for the trial
* Uncontrolled peripheral neuropathy (more than grade 2)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-11-10 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Evaluate MRI good response rate after the total neoadjuvant treatment | 16-20 weeks after SCRT
  Good response rate is defined as the proportion of patients who reached mrTRG 1 or 2 and the absence of remote disease in the reevaluation period, with the denominator being the total number of patients who started total neoadjuvant treatment.

SECONDARY OUTCOMES:
Disease-free survival in 3 years | 3 years
  defined as the time from the date of MRI of the pelvis of the reassessment period to relapse, death or last contact date.
Overall survival | 3 years
  defined as the time from the date of the induction chemotherapy until the death or date of last contact
Describe the safety and tolerability of total neoadjuvant treatment. | 1 year
  Incidence of adverse events (AEs), serious AEs, deaths and laboratory abnormalities in participants who received at least one dose of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Juliana Souza, Principal Investigator — Instituto Nacional de Cancer, Brazil
Locations (1):
- INCA- Instituto Nacional de Câncer, Rio de Janeiro, Brazil